CLINICAL TRIAL: NCT06182306
Title: Prospective Evaluation of AI R&D Tool for Patient Stratification - Mechanism of Action Evaluation in Triple Negative Breast Cancer (PEAR-MET)
Brief Title: Prospective Evaluation of AI R&D Tool for Patient Stratification - MoA Evaluation in Triple Negative Breast Cancer (PEAR-MET)
Acronym: PEAR-MET
Status: Recruiting | Type: Observational
Sponsor: Ourotech, Inc. (Industry)
Collaborators: Guys' and St. Thomas Hospital (Unknown); Barts & The London NHS Trust (Other); Imperial College Healthcare NHS Trust (Other); Nottingham University Hospitals Trust (Unknown); Hampshire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PEAR-MET
Record Dates: First submitted 2023-12-08; First posted 2023-12-26 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
Keywords: computer vision; cell culture; microtumor; functional testing; predictive biomarker
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor cores and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trial Cohort: Patients with advanced or metastatic triple negative breast cancer, due to start a new line of systemic therapy (targeted drug or immunotherapy)
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Patients undergo a biopsy from a lesion, and give 40ml of blood

SUMMARY:
Pear Bio has developed an organ-on-a-chip device together with a computer vision pipeline through which the response of an individual patient's tumor to different systemic therapy regimens can be tested simultaneously ex vivo. This study will recruit patients with advanced or metastatic triple negative breast cancer who are due to start a clinically-indicated new line of therapy.

The oncologist will be blinded to the response on the Pear Bio tool (the assay will be run in parallel with the patient's treatment). The primary objective of this study is to establish the sensitivity and specificity of Pear Bio's test against patient outcomes (response, progression-free survival, overall survival)

DETAILED DESCRIPTION:
This is a UK-based observational study that aims to discover novel predictive biomarkers with the potential to guide treatment decision making and prolong PFS and OS in patients with advanced TNBC. Patients will undergo a mandatory, study-specific core needle biopsy or fine needle aspiration of the breast tumour or metastasis before commencing their next line of therapy. The research sample will be run on Pear Bio's test whilst the patient receives therapy as per their physician's choice. This study will not use Pear Bio's tool to inform the choice of treatment, with the treating oncologist being blinded to the test results. Treatment response data will be collected at multiple timepoints to conduct analyses on the study's secondary and tertiary objectives.

Fresh tissue resections that arrive at Pear Bio's lab will undergo processing, cell culture and various drug dosing and omics assays (depending on extracted cell numbers). Tumour samples will be processed using a cell isolation kit to retrieve a viable single-cell suspension. A minimum of 100,000 cells (10,000 viable cells per chip) will be used for staining with live and dead cell-tracking dyes. In parallel, blood vials will be processed for PBMCs and further effector cell extraction (flow cytometry, Dynabeads, etc). The remaining cells will be used for sequencing (DNA/RNA), fixed for immunofluorescence characterisation of biomarkers/receptor status or used for further omics assays (if cell numbers allow). This may include tumour mutational burden and microsatellite instability testing.

The stained cells will be cultured in a biomimetic hydrogel within Pear Bio's organ-on-a-chip to provide a physiological 3D environment for drug dosing experiments. Using a microfluidic device, samples in each chip will be exposed to approved therapies (either as monotherapy or combination therapies, as outlined below) over multiple days.

In parallel, PBMCs will be extracted from whole blood, characterised and sorted via flow cytometry and fluorescence-activated cell sorting (FACS) or magnetic beads selection. Cells of interest (e.g. CD8+ T cells) will be used for culture in Pear Bio's chips jointly with cells isolated from the matched tumour sample. To test immunotherapies, tumour cells will be co-cultured with immune cells in a modified organ-on-a-chip architecture. Chips receiving immunotherapies may be tested for tumour mutational burden and/or microsatellite instability.

Confocal microscopy will be conducted daily to collect 3D image data of the cells and track their position and behaviour over time. At the end of the assay, the 3D cell cultures will be fixed for further 3D immunofluorescence analyses or used for embedding, sectioning and assessment of spatial transcriptomics. For targeted therapies, RNAseq, IF and other omics data will be integrated to confirm drug MoA and identify other potential therapeutic targets. Concurrently, 3D image data is processed through a computer vision pipeline to measure functional metrics of the ex vivo 3D cell cultures, including cell viability, cell culture width and cell migration, both at a bulk tumour level and at a single-cell resolution. For immunotherapies, additional metrics such as immune cell infiltration and immune cell killing will be recorded. A patient report is then generated to outline an individual patient sample's response to each therapy tested.

ELIGIBILITY:
Inclusion criteria

1. Able to give written informed consent prior to admission to this study.
2. Female or male aged ≥18 years.
3. Histologically confirmed primary breast cancer which is triple-negative by the most recent ASCO/College of American Pathologists (CAP) guidelines.

   Stage 4 or locally advanced breast cancer planned for first line systemic therapy, or has received prior lines of systemic therapy and is due to undergo another line of systemic therapy.
4. Willing and able to undergo a mandatory additional core needle biopsy (minimum 2 cores) or equivalent fine needle aspiration from the primary breast mass or a metastasis prior to starting the subsequent line of systemic therapy.
5. Willing and able to undergo a mandatory procedure to collect 40 mL of blood.

Exclusion criteria

1. Tumours not confirmed as triple negative breast cancer.
2. Early stage TNBC.
3. Patients with TNBC that do not intend to receive systemic therapy.
4. Patients who have already commenced systemic therapy with no plans of changing the systemic therapy after the collection of the core needle biopsy or fine needle aspirate sample.
5. Patients who are due to receive experimental therapies that are not included in the study protocol.
6. Haemoglobin levels below 80g/L prior to research sample collection.
7. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced or metastatic triple negative breast cancer, due to start a new line of therapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Establish a functional dose of each commonly used FDA approved therapeutic/combination | 6 months
  To conduct dose-response analysis for each commonly used FDA approved therapy, or combination of therapies, to establish the correct dose in the Pear Bio system

SECONDARY OUTCOMES:
ORR prediction accuracy | 3 months
  The performance (sensitivity, specificity, PPV and NPV) of Pear image-based biomarkers are established against patients' overall response rate (ORR) as defined by RECIST 1.1 guidelines
PFS prediction accuracy | 12-24 months
  The performance of Pear image-based biomarkers are established against patients' progression-free survival at 6, 12 and 24 months (evaluated by imaging).
OS prediction accuracy | 2 years
  The performance of Pear image-based biomarkers are established against patients' overall survival at 6, 12 and 24 months (evaluated by imaging).

OTHER OUTCOMES:
Culture success rate | 4 days
  The percentage of patient samples successfully arriving at central lab with >100k live cells isolated and maintaining 70% cell viability after 4 days in culture with no treatment
Assess the correlation of various "omic" biomarkers to patient PFS, ORR and/or OS | 2 years
  The relationship between DNA, RNA and protein levels and patient outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Sheeba Irshad, MD PhD, Principal Investigator — King's College London
Locations (3):
- United Kingdom (3):
  - Imperial College Healthcare NHS Trust, London
  - Barts Hospital NHS Trust, London
  - Guys and St. Thomas Hospital NHS Trust, London

IPD SHARING:
Plan to Share IPD: No
Pseudonymised data will be shared between study sites, such as treatment and outcome data for each patient. No publication will be made revealing individual patient data; only group-level data will be published.

REFERENCES:
- Available data/document: Study Protocol — https://www.pearbio.com/pearmet — Company website with background and information and links to protocol, etc.